CLINICAL TRIAL: NCT03606928
Title: Modified FLOT Chemotherapy as First-line Treatment in Advanced or Metastatic Gastric Cancer
Brief Title: mFLOT Chemotherapy as First-line Treatment in GC
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Jun Zhang, Chief, Department of Oncology, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: mFLOT-GC
Record Dates: First submitted 2018-07-22; First posted 2018-07-31 (Actual); Last update posted 2020-03-20 (Actual); Status verified 2020-03

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Docetaxel; Oxaliplatin; Fluorouracil; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- modified FLOT (Experimental): modified FLOT Docetaxel 40mg/m2 ivgtt day 1 over 1 hour Oxaliplatin 65mg/m2 ivgtt day 1 over 2hours Dose escalation will be performed. Leucovorin 200mg/m2 ivgtt day 1 over 2 hours 5-FU 2200mg/m2 civ over 24 hours
  Interventions: Drug: docetaxel, oxaliplatin, 5-FU, leucovorin

INTERVENTIONS:
Drug: docetaxel, oxaliplatin, 5-FU, leucovorin — This is a single-arm study with all patients receiving mFLOT chemotherapy.

SUMMARY:
A single center phase 1b/2 trail to identified suitable dosage and its efficacy of modified FLOT regime in Chinese gastric cancer patients. This trial is designed to identified recommended phase II dose (RP2D) of modified FLOT in Chinese patients, and to evaluate the efficacy of modified FLOT regime as first-line for advanced or metastatic gastric cancer.

This trial is in 2 stages: the first stage will establish the maximum tolerated dose (MTD) and RP2D of docetaxel and oxaliplatin in FLOT regime. In the second stage, the efficacy of modified FLOT will be assessed by response rate.

DETAILED DESCRIPTION:
The RP2D of FLOT regime will be established with a standard 3+3 design, starting with the dose of 40mg/m2 docetaxel (dose level 1) and 65mg/m2 oxaliplatin (dose level 1). The plan of dose escalation will be found in following table. Chemotherapy will be administered two-weekly (maximum 12 cycles) until progression of disease, intolerable toxicity or withdraw of patients.

ELIGIBILITY:
Inclusion Criteria:

1. Male/female patients aged from 18 to 75 years.
2. Histologically confirmed gastric adenocarcinoma.
3. Gastric tumors should be treatment naïve unresectable or metastatic disease, or recurrence over 6 months after finish of adjuvant chemotherapy.
4. At least one measurable lesion should be confirmed by imaging examination.
5. ECOG performance status 0 or 1
6. Adequate bone marrow function:

   Absolute neutrophil count (ANC) ≥1.5x109/L White blood count ≥3.5x109/L Platelets ≥80x109/L Hemoglobin (Hb) ≥90g/L (can be post-transfusion)
7. Adequate renal function: Creatinine Clearance of >50ml/min
8. Adequate liver function:

Serum bilirubin <22 umol/L ALT/AST ≤2.5x ULN, for patient with liver metastasis ALT/AST ≤5x ULN 10. Adequate coagulation profile International Normalised Ratio (INR) < 1.5 Activated Prothrombin Time (APTT) < 1.5xULN 11. Without brain metastasis and peripheral nerve diseases 12. Willingness and ability to comply with the protocol for the duration of the study including scheduled visits, examinations, investigations and treatment plans with informed consent form.

Exclusion Criteria:

1. With second primary malignant diseases
2. Any contraindication or known hypersensitivity reaction to any of the study drugs, or components of leucovorin, oxaliplatin, 5-FU or docetaxel
3. With uncontrollable complications
4. Inadequate organ function
5. Pregnancy or of child bearing potential.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-11-09 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose and recommended phase II dose of modified FLOT regime | 36 months
Objective response rate | 36 months

SECONDARY OUTCOMES:
Overall survival | 36 months
Progression free survival | 36 months
Safety: adverse events as assessed by CTCAE v4.0 | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Jun Zhang, MD & Ph. D, Principal Investigator — Ruijin Hospital
Locations (1):
- Department of Oncology, Ruijin Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No
We have no plan to make individual participant data (IPD) available to other researchers.

DOCUMENTS (2):
  • Study Protocol (2018-05-02): https://cdn.clinicaltrials.gov/large-docs/28/NCT03606928/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-02): https://cdn.clinicaltrials.gov/large-docs/28/NCT03606928/SAP_001.pdf